CLINICAL TRIAL: NCT07056491
Title: Serum REST4 as a Predictive Biomarker for Abdominal Aortic Aneurysm Progression
Brief Title: REST4-AAA Registry
Acronym: REST4 Registry
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REST4-AAA
Record Dates: First submitted 2025-06-19; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study need to retain processed serum samples from participants to isolate exosome and quantify the REST4 mRNA level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mRNA level of REST4 in serum; — 1. mRNA level of REST4 in serum The mRNA expression level of REST4 was measured in serum-derived exosomes using RT-qPCR at the time of patient enrollment.
  2. Computed tomography angiography (CTA) Baseline maximum internal diameter of the abdominal aortic aneurysm (AAA) was determined by CTA at enrollment. During follow-up, CTA was performed to assess the increase in maximum AAA diameter.

SUMMARY:
This prospective observational study aims to investigate whether serum REST4 concentration can serve as a quantitative indicator correlated with abdominal aortic aneurysm (AAA) diameter and a predictive biomarker for AAA progression and rupture risk. Emerging evidence suggests that REST4, a splice variant of the RE-1 Silencing Transcription Factor (REST), is upregulated in vascular smooth muscle cells during AAA pathogenesis and may be released into circulation via exosomes. The study will enroll patients with asymptomatic AAA (diameter between 39-49 mm) and measure baseline serum REST4 levels, analyzing their association with morphological severity (maximum aortic diameter) and clinical outcomes (aneurysm growth rate, rupture and related mortality) through a 5-year follow-up period.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is a life-threatening vascular disease characterized by progressive dilation of the abdominal aorta, ultimately leading to catastrophic rupture with high mortality. Currently, clinical management relies mainly on aneurysm diameter for risk assessment, lacking reliable biomarkers to predict disease progression or rupture risk. Emerging evidence highlights the critical role of vascular smooth muscle cell (VSMC) phenotypic switching in AAA pathogenesis. Preliminary research has identified that RE-1 Silencing Transcription Factor (REST) in VSMC undergoes alternative splicing in AAA tissues, resulting in predominant expression of its splice variant REST4 and downregulation of full-length REST. This molecular shift triggers STAT1 activation, promoting synthetic VSMC transformation.

The study hypothesizes that synthetic VSMC in AAA lesions secrete REST4 into circulation via exosomes, making serum REST4 a potential dual-parameter biomarker that quantitatively correlates with aneurysm diameter (morphological severity) and predicts disease progression and rupture risk.

This prospective observational study will systematically evaluate asymptomatic AAA patients (39-49 mm diameter) to first determine the relationship between serum REST4 levels and maximum aortic diameter. Subsequently, through 5-year follow-up, the investigators will assess the prognostic capacity of serum REST4 concentration for predicting annual aneurysm growth rates, rupture incidence, and aneurysm-specific mortality.

Validation of correlation between serum REST4 concentration and AAA progression could transform current AAA surveillance approaches by integrating molecular profiling with traditional anatomical monitoring, enabling more precise risk stratification and personalized clinical management to ultimately improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an infrarenal AAA with a maximum diameter of 39-49 mm;
2. Han nationality;
3. Between 50 years or more, no gender limit;
4. No mental illness;
5. Subjects voluntarily participate in this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Previous infrarenal aortic surgery;
2. Planned major surgery;
3. Known aortic dissection;
4. Have received any other clinical trial treatment within 1 year;
5. Systemic treatment with corticosteroids or other systemic immunomodulatory therapy;
6. Severe infections, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.;
7. Known or suspected inherited connective tissue disorder;
8. Known or suspected prostate cancer;
9. Calculated creatinine clearance of less than 30 ml/min;
10. Known significant liver disease;
11. Known human immunodeficiency virus infection at the time of screening；
12. Serious concomitant illness associated with life expectancy of less than 2 years；
13. Any other significant and unstable condition that could limit compliance with the trial protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With an Abdominal Aortic Aneurysm of 39-49 mm in Diameter.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Serum REST4 Level | Baseline
  Quantification of serum REST4 mRNA levels in enrolled patients using RT-qPCR method
Maximal diameter of abdominal aorta | Baseline
  Measurement of maximal diameter of infrarenal abdominal aorta from leading edge adventitia at the anterior wall to leading edge adventitia at the posterior wall by computed tomography angiography
Change in abdominal aortic diameter | 5 years
  Measurement of maximal diameter of infrarenal abdominal aorta from leading edge adventitia at the anterior wall to leading edge adventitia at the posterior wall by computed tomography angiography during 5-year follow-up period.

SECONDARY OUTCOMES:
Rates of AAA repair/rupture | 5 years
  Calculate the incidence of AAA repair/rupture
Mortality | 5 years
  Calculate the mortality due to AAA rupture

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided